CLINICAL TRIAL: NCT04279483
Title: Geo Smoking Study and Neural and Geospatial Examination of Smokers' Exposure to Retail Environments
Brief Title: GeoScan and Remote Geo Smoking Study: Neural and Behavioral Correlates of Smokers' Exposure to Retail Environments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New York University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 822815, 850796; 1R01CA229305-01A1 (NIH)
Record Dates: First submitted 2020-02-14; First posted 2020-02-21 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Smoking, Tobacco; Smoking; Smoking, Cigarette
Keywords: smoking; smoker; tobacco; cigarette; cigarettes; Philadelphia; healthy
MeSH Terms: conditions — Tobacco Smoking; Smoking; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Random assignment of retail environment (tobacco retailer, non-tobacco retailer, control [no store]) to visit 5 times per week during the 4-week intervention period
Who Masked: Investigator
Masking Description: Investigator will not know the condition assignment of individual participants unless reassessment is triggered by the stopping rule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tobacco Retailer Group (Experimental): Participants visit a tobacco retailer 5 times per week during the 4-week (20 store visits total) intervention period
  Interventions: Behavioral: Tobacco retailer
- Non-tobacco Retailer Group (Experimental): Participants visit a non-tobacco retailer 5 times per week during the 4-week (20 store visits total) intervention period
  Interventions: Behavioral: Non-tobacco retailer
- Control (No Intervention): Participants are not asked to alter their behavior during the 4-week (0 store visits) intervention period

INTERVENTIONS:
Behavioral: Tobacco retailer — Assigned to make a small (~$3.00) purchase from a tobacco retail store(s) using a study-provided debit card during each retail environment visit
  Arms: Tobacco Retailer Group
Behavioral: Non-tobacco retailer — Assigned to make a small (~$3.00) purchase from a store that does not sell tobacco (non-tobacco retailer) using a study-provided debit card during each retail environment visit.
  Arms: Non-tobacco Retailer Group

SUMMARY:
The purpose of the study is to learn more about the relationships between the brain, behavior, and natural daily exposure to particular environments, including the places where smokers regularly spend time and specific retail outlets.

DETAILED DESCRIPTION:
Individual participation in this study will take place over a period of approximately 2 months. During (approximately) 6 weeks of the active study period, the participant will be asked to share their geolocation information, complete either (a) 3 online sessions (for all participants in 850796) and an optional fMRI scan (for a subset of protocol 850796) or (b) 3 in-person visits (2 of which involve getting fMRI brain scans, for protocol 822815), and complete short surveys and repeated tasks (e.g., responding to Ecological Momentary Assessment [EMA], using study-provided funds to make small purchases from a specified retail environment) in the weeks between visits.

ELIGIBILITY:
Inclusion criteria:

* Be between the ages of 21-65
* Smoke at least 5 cigarettes a day for the past 6 months
* Own an iPhone or Android smartphone that can be used on a daily basis
* Plan to be in PA, DE, or NJ (for the remote cohort) or the Philadelphia metropolitan area (for the fMRI cohort) for the next 3 months, with the exception of short periods of absence (no longer than 3 consecutive days and no more than 10 days in total)
* Read and speak English fluently
* Fully vaccinated against COVID-19

Smoking exclusion criteria:

* Current enrollment or plans to enroll in a smoking cessation program in the next 3 months
* Plan to use nicotine substitutes or smoking cessation treatments in the next 3 months
* Urine cotinine test at Session 1 indicates a non-smoker level of cotinine

General exclusion criteria:

* Pregnancy
* Inability or refusal to install Google Maps or LifeData applications on mobile phone
* Inability or refusal to upload Google Timeline data after receiving instructions and guidance from a researcher
* Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.
* Any physical or visual impairment that may prevent the individual from using a computer keyboard or completing any study tasks.
* During the first two weeks of the study, failure to complete the study tasks (e.g., response to at least 75% of the brief EMA survey questions).
* The phones of potential participants will be assessed by trained recruiters either during in-person recruiting or during a phone call used to invite eligible participants who filled out the online screening survey for the first appointment. Specifically, recruiters will assess whether phones' functionality allows easy reception and sending of text messages, the use of the geolocation tracking and LifeData applications, whether potential participants have an existing Google account (created prior to Jan 2024), and whether phones have an adequate battery life to allow participants to fulfill study requirements.
* Any medical condition or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.

Drug & fMRI exclusion criteria (fMRI cohort only - 822815 participants and fMRI subset of 850796 participants):

* Currently or recently (within the last 5 years) receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana, or stimulants). Treatment of substance use disorders that occurred greater than 5 years prior to study participation is acceptable if participants are in stable condition
* Report consuming any of the following drugs within the past two weeks or indicate plans to do so within the coming 6 weeks during the initial recruitment call: Benzodiazepines, Amphetamines, Methamphetamines, Cocaine, MDMA, Methadone, Barbiturates, PCP, Heroin, Oxycodone, Opiates (e.g., morphine, heroin), Buprenorphine.
* Test positive for any of the above drugs at Appointment 1 (822815) or at the scan appointment (850796)
* Schizophrenia or psychosis, regardless of treatment status
* History of stroke or other neurological disorder likely to affect cognition
* For 850796, history of seizures, brain tumor, penetrative head trauma that cracks the skull
* Psychiatric hospitalization within the past year

MRI exclusion criteria:

* For 850796, history of problems in previous MRI that are likely to occur again
* For 822815, left-handedness
* Propensity to experience claustrophobia
* Ferromagnetic metal in the body, including anything that might set off a metal detector. Examples include bullet shrapnel, metal shavings (e.g., from welding without protection), or any implant that may be attracted to or damaged by magnets. Dental fillings are generally acceptable.
* Metal in the body of an unverifiable origin
* Non-removable piercings
* Non-removable retainers or other dental work not compatible with fMRI.
* Any orthopedic implant above the neck
* Due to constraints of the fMRI scanner, participants whose weight exceeds 350 pounds also will be excluded
* For 850796, scan must be scheduled within 6 months after completing the third Online Session

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Falk, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
* The final data set will include data from 310 subjects in PA, NJ, or DE. Data (collected via questionnaires, urine cotinine assessments, and smartphone applications) will include measures concerned with health behaviors, individuals' geospatial distance from nearby tobacco retail outlets, and personality and individual differences. 822815 and the fMRI subset of 850796 will include data from the brain imaging scan(s). 822815 will also include saliva cotinine assessments conducted during 2 of the 3 in-person sessions.
  * Final research data, with all identity-related information deleted and in consultation with the relevant IRBs, will be made available to scientists who are approved by the study team for collaborative research with members of the study team. Data will be shared in spreadsheet format for all non-imaging data and in NIFTI format for fMRI data. Unthresholded statistical maps for the fMRI data will be made available to researchers through a secure file-sharing interface.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available within six months following publication of the study's primary results. Data will remain available for a minimum of three years following the closeout of the grant.
Access Criteria: * Data will be made available to scientists who are approved by the study team for collaborative research with members of the study team.
  * Qualified investigators who wish to access the study materials will be able to complete a form on the main project website on GitHub (https://github.com/cnlab), which describes the proposed study and delineates the data specifics of data use. The requests will be reviewed and approved by the investigators. The requested research data files will be accompanied by a description of variables and how they were collected. We will also share protocols relevant to data collection procedures, as useful and in consultation with other interested researchers.
  * Study tasks and code to reproduce analyses will be made available on the Falk lab GitHub account (https://github.com/cnlab)
  * Statistical Analysis Plans will be available in the form of pre-registrations on the Open Science Framework site (https://osf.io).
URL: https://docs.google.com/document/d/1UkubuRug0gY8DEkTiB75fgcJuxdwlBZtmeY4qrUfog4/edit?usp=sharing

REFERENCES:
- [Background] Wakefield MA, Terry-McElrath YM, Chaloupka FJ, Barker DC, Slater SJ, Clark PI, Giovino GA. Tobacco industry marketing at point of purchase after the 1998 MSA billboard advertising ban. Am J Public Health. 2002 Jun;92(6):937-40. doi: 10.2105/ajph.92.6.937. No abstract available. PMID 12036782
- [Background] Henriksen L. Comprehensive tobacco marketing restrictions: promotion, packaging, price and place. Tob Control. 2012 Mar;21(2):147-53. doi: 10.1136/tobaccocontrol-2011-050416. PMID 22345238
- [Background] Henriksen L, Ribisl KM, Rogers T, Moreland-Russell S, Barker DM, Sarris Esquivel N, Loomis B, Crew E, Combs T. Standardized Tobacco Assessment for Retail Settings (STARS): dissemination and implementation research. Tob Control. 2016 Oct;25(Suppl 1):i67-i74. doi: 10.1136/tobaccocontrol-2016-053076. PMID 27697950
- [Background] Feld AL, Johnson TO, Byerly KW, Ribisl KM. How to Conduct Store Observations of Tobacco Marketing and Products. Prev Chronic Dis. 2016 Feb 18;13:E25. doi: 10.5888/pcd13.150504. PMID 26890408
- [Background] Li L, Borland R, Fong GT, Thrasher JF, Hammond D, Cummings KM. Impact of point-of-sale tobacco display bans: findings from the International Tobacco Control Four Country Survey. Health Educ Res. 2013 Oct;28(5):898-910. doi: 10.1093/her/cyt058. Epub 2013 May 2. PMID 23640986
- [Background] Kirchner TR, Cantrell J, Anesetti-Rothermel A, Ganz O, Vallone DM, Abrams DB. Geospatial exposure to point-of-sale tobacco: real-time craving and smoking-cessation outcomes. Am J Prev Med. 2013 Oct;45(4):379-85. doi: 10.1016/j.amepre.2013.05.016. PMID 24050412
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Engelmann JM, Versace F, Robinson JD, Minnix JA, Lam CY, Cui Y, Brown VL, Cinciripini PM. Neural substrates of smoking cue reactivity: a meta-analysis of fMRI studies. Neuroimage. 2012 Mar;60(1):252-62. doi: 10.1016/j.neuroimage.2011.12.024. Epub 2011 Dec 21. PMID 22206965
- [Background] McClernon FJ, Hiott FB, Huettel SA, Rose JE. Abstinence-induced changes in self-report craving correlate with event-related FMRI responses to smoking cues. Neuropsychopharmacology. 2005 Oct;30(10):1940-7. doi: 10.1038/sj.npp.1300780. PMID 15920499
- [Background] McClernon FJ, Conklin CA, Kozink RV, Adcock RA, Sweitzer MM, Addicott MA, Chou YH, Chen NK, Hallyburton MB, DeVito AM. Hippocampal and Insular Response to Smoking-Related Environments: Neuroimaging Evidence for Drug-Context Effects in Nicotine Dependence. Neuropsychopharmacology. 2016 Feb;41(3):877-85. doi: 10.1038/npp.2015.214. Epub 2015 Jul 16. PMID 26179147
- [Background] Henriksen L, Schleicher NC, Feighery EC, Fortmann SP. A longitudinal study of exposure to retail cigarette advertising and smoking initiation. Pediatrics. 2010 Aug;126(2):232-8. doi: 10.1542/peds.2009-3021. Epub 2010 Jul 19. PMID 20643725
- [Background] Robertson L, McGee R, Marsh L, Hoek J. A systematic review on the impact of point-of-sale tobacco promotion on smoking. Nicotine Tob Res. 2015 Jan;17(1):2-17. doi: 10.1093/ntr/ntu168. Epub 2014 Aug 30. PMID 25173775
- [Background] Burton S, Clark L, Jackson K. The association between seeing retail displays of tobacco and tobacco smoking and purchase: findings from a diary-style survey. Addiction. 2012 Jan;107(1):169-75. doi: 10.1111/j.1360-0443.2011.03584.x. Epub 2011 Oct 7. PMID 21777322
- [Background] Carter OB, Phan T, Mills BW. Impact of a point-of-sale tobacco display ban on smokers' spontaneous purchases: comparisons from postpurchase interviews before and after the ban in Western Australia. Tob Control. 2015 Mar;24(e1):e81-6. doi: 10.1136/tobaccocontrol-2013-050991. Epub 2013 Dec 23. PMID 24365702
- [Background] Carter OB, Mills BW, Donovan RJ. The effect of retail cigarette pack displays on unplanned purchases: results from immediate postpurchase interviews. Tob Control. 2009 Jun;18(3):218-21. doi: 10.1136/tc.2008.027870. Epub 2009 Mar 4. PMID 19264731
- [Background] Wakefield M, Germain D, Henriksen L. The effect of retail cigarette pack displays on impulse purchase. Addiction. 2008 Feb;103(2):322-8. doi: 10.1111/j.1360-0443.2007.02062.x. Epub 2007 Nov 27. PMID 18042190
- [Background] Siahpush M, Shaikh RA, Smith D, Hyland A, Cummings KM, Kessler AS, Dodd MD, Carlson L, Meza J, Wakefield M. The Association of Exposure to Point-of-Sale Tobacco Marketing with Quit Attempt and Quit Success: Results from a Prospective Study of Smokers in the United States. Int J Environ Res Public Health. 2016 Feb 6;13(2):203. doi: 10.3390/ijerph13020203. PMID 26861379
- [Background] Siahpush M, Shaikh RA, Cummings KM, Hyland A, Dodd M, Carlson L, Kessler AS, Meza J, Wan N, Wakefield M. The association of point-of-sale cigarette marketing with cravings to smoke: results from a cross-sectional population-based study. Tob Control. 2016 Jul;25(4):402-5. doi: 10.1136/tobaccocontrol-2015-052253. Epub 2015 May 29. PMID 26024797
- [Background] Henriksen L, Feighery EC, Schleicher NC, Cowling DW, Kline RS, Fortmann SP. Is adolescent smoking related to the density and proximity of tobacco outlets and retail cigarette advertising near schools? Prev Med. 2008 Aug;47(2):210-4. doi: 10.1016/j.ypmed.2008.04.008. Epub 2008 Apr 29. PMID 18544462
- [Background] Lipperman-Kreda S, Mair C, Grube JW, Friend KB, Jackson P, Watson D. Density and proximity of tobacco outlets to homes and schools: relations with youth cigarette smoking. Prev Sci. 2014 Oct;15(5):738-44. doi: 10.1007/s11121-013-0442-2. PMID 24254336
- [Background] Pearce J, Hiscock R, Moon G, Barnett R. The neighbourhood effects of geographical access to tobacco retailers on individual smoking behaviour. J Epidemiol Community Health. 2009 Jan;63(1):69-77. doi: 10.1136/jech.2007.070656. Epub 2008 Jul 15. PMID 18628269
- [Background] Cantrell J, Anesetti-Rothermel A, Pearson JL, Xiao H, Vallone D, Kirchner TR. The impact of the tobacco retail outlet environment on adult cessation and differences by neighborhood poverty. Addiction. 2015 Jan;110(1):152-61. doi: 10.1111/add.12718. Epub 2014 Nov 7. PMID 25171184
- [Background] Reitzel LR, Cromley EK, Li Y, Cao Y, Dela Mater R, Mazas CA, Cofta-Woerpel L, Cinciripini PM, Wetter DW. The effect of tobacco outlet density and proximity on smoking cessation. Am J Public Health. 2011 Feb;101(2):315-20. doi: 10.2105/AJPH.2010.191676. Epub 2010 Dec 16. PMID 21164089
- [Background] Chaiton M, Mecredy G, Rehm J, Samokhvalov AV. Tobacco retail availability and smoking behaviours among patients seeking treatment at a nicotine dependence treatment clinic. Tob Induc Dis. 2014 Dec 2;12(1):19. doi: 10.1186/1617-9625-12-19. eCollection 2014. PMID 25745380
- [Background] Kim AE, Nonnemaker JM, Loomis BR, Shafer PR, Shaikh A, Hill E, Holloway JW, Farrelly MC. Influence of point-of-sale tobacco displays and graphic health warning signs on adults: evidence from a virtual store experimental study. Am J Public Health. 2014 May;104(5):888-95. doi: 10.2105/AJPH.2013.301723. Epub 2014 Mar 13. PMID 24625149
- [Background] Hubbeling HG, Frank DM, Hexner EO. Myelofibrosis 2012: it's complicated. Ther Adv Hematol. 2012 Jun;3(3):131-46. doi: 10.1177/2040620712437754. PMID 23556120
- [Background] Shiffman S. Ecological momentary assessment (EMA) in studies of substance use. Psychol Assess. 2009 Dec;21(4):486-97. doi: 10.1037/a0017074. PMID 19947783
- [Background] Berkman ET, Dickenson J, Falk EB, Lieberman MD. Using SMS text messaging to assess moderators of smoking reduction: Validating a new tool for ecological measurement of health behaviors. Health Psychol. 2011 Mar;30(2):186-94. doi: 10.1037/a0022201. PMID 21401252
- [Background] Konrath S, Falk E, Fuhrel-Forbis A, Liu M, Swain J, Tolman R, Cunningham R, Walton M. Can Text Messages Increase Empathy and Prosocial Behavior? The Development and Initial Validation of Text to Connect. PLoS One. 2015 Sep 10;10(9):e0137585. doi: 10.1371/journal.pone.0137585. eCollection 2015. PMID 26356504
- [Background] Carter BL, Tiffany ST. Meta-analysis of cue-reactivity in addiction research. Addiction. 1999 Mar;94(3):327-40. PMID 10605857
- [Background] Tiffany ST. A cognitive model of drug urges and drug-use behavior: role of automatic and nonautomatic processes. Psychol Rev. 1990 Apr;97(2):147-68. doi: 10.1037/0033-295x.97.2.147. PMID 2186423
- [Background] Zubieta JK, Heitzeg MM, Xu Y, Koeppe RA, Ni L, Guthrie S, Domino EF. Regional cerebral blood flow responses to smoking in tobacco smokers after overnight abstinence. Am J Psychiatry. 2005 Mar;162(3):567-77. doi: 10.1176/appi.ajp.162.3.567. PMID 15741475
- [Background] Brody AL, Mandelkern MA, London ED, Childress AR, Lee GS, Bota RG, Ho ML, Saxena S, Baxter LR Jr, Madsen D, Jarvik ME. Brain metabolic changes during cigarette craving. Arch Gen Psychiatry. 2002 Dec;59(12):1162-72. doi: 10.1001/archpsyc.59.12.1162. PMID 12470133
- [Background] Shiffman S, Dunbar M, Kirchner T, Li X, Tindle H, Anderson S, Scholl S. Smoker reactivity to cues: effects on craving and on smoking behavior. J Abnorm Psychol. 2013 Feb;122(1):264-80. doi: 10.1037/a0028339. Epub 2012 Jun 18. PMID 22708884
- [Background] Conklin CA, Perkins KA, Robin N, McClernon FJ, Salkeld RP. Bringing the real world into the laboratory: personal smoking and nonsmoking environments. Drug Alcohol Depend. 2010 Sep 1;111(1-2):58-63. doi: 10.1016/j.drugalcdep.2010.03.017. Epub 2010 May 26. PMID 20510552
- [Background] Japuntich SJ, Piper ME, Leventhal AM, Bolt DM, Baker TB. The effect of five smoking cessation pharmacotherapies on smoking cessation milestones. J Consult Clin Psychol. 2011 Feb;79(1):34-42. doi: 10.1037/a0022154. PMID 21261432
- [Background] Wang AL, Ruparel K, Loughead JW, Strasser AA, Blady SJ, Lynch KG, Romer D, Cappella JN, Lerman C, Langleben DD. Content matters: neuroimaging investigation of brain and behavioral impact of televised anti-tobacco public service announcements. J Neurosci. 2013 Apr 24;33(17):7420-7. doi: 10.1523/JNEUROSCI.3840-12.2013. PMID 23616548
- [Background] Falk EB, Berkman ET, Lieberman MD. From neural responses to population behavior: neural focus group predicts population-level media effects. Psychol Sci. 2012 May 1;23(5):439-45. doi: 10.1177/0956797611434964. Epub 2012 Apr 17. PMID 22510393
- [Background] Falk EB, O'Donnell MB, Tompson S, Gonzalez R, Dal Cin S, Strecher V, Cummings KM, An L. Functional brain imaging predicts public health campaign success. Soc Cogn Affect Neurosci. 2016 Feb;11(2):204-14. doi: 10.1093/scan/nsv108. Epub 2015 Sep 23. PMID 26400858
- [Background] Pegors TK, Tompson S, O'Donnell MB, Falk EB. Predicting behavior change from persuasive messages using neural representational similarity and social network analyses. Neuroimage. 2017 Aug 15;157:118-128. doi: 10.1016/j.neuroimage.2017.05.063. Epub 2017 May 31. PMID 28578131
- [Background] Cooper N, Bassett DS, Falk EB. Coherent activity between brain regions that code for value is linked to the malleability of human behavior. Sci Rep. 2017 Feb 27;7:43250. doi: 10.1038/srep43250. PMID 28240271
- [Background] Green AE, Mays D, Falk EB, Vallone D, Gallagher N, Richardson A, Tercyak KP, Abrams DB, Niaura RS. Young Adult Smokers' Neural Response to Graphic Cigarette Warning Labels. Addict Behav Rep. 2016 Jun 1;3:28-32. doi: 10.1016/j.abrep.2016.02.001. PMID 27019865
- [Background] Cooper N, Tompson S, O'Donnell MB, Falk EB. Brain Activity in Self- and Value-Related Regions in Response to Online Antismoking Messages Predicts Behavior Change. J Media Psychol. 2015;27:93-109. doi: 10.1027/1864-1105/a000146. Epub 2015 Sep 15. PMID 29057013
- [Background] Vezich IS, Katzman PL, Ames DL, Falk EB, Lieberman MD. Modulating the neural bases of persuasion: why/how, gain/loss, and users/non-users. Soc Cogn Affect Neurosci. 2017 Feb 1;12(2):283-297. doi: 10.1093/scan/nsw113. PMID 27521303
- [Background] Falk EB, Berkman ET, Whalen D, Lieberman MD. Neural activity during health messaging predicts reductions in smoking above and beyond self-report. Health Psychol. 2011 Mar;30(2):177-85. doi: 10.1037/a0022259. PMID 21261410
- [Background] Falk EB, Berkman ET, Mann T, Harrison B, Lieberman MD. Predicting persuasion-induced behavior change from the brain. J Neurosci. 2010 Jun 23;30(25):8421-4. doi: 10.1523/JNEUROSCI.0063-10.2010. PMID 20573889
- [Background] Huskey R, Mangus JM, Turner BO, Weber R. The persuasion network is modulated by drug-use risk and predicts anti-drug message effectiveness. Soc Cogn Affect Neurosci. 2017 Dec 1;12(12):1902-1915. doi: 10.1093/scan/nsx126. PMID 29140500
- [Background] Falk EB, O'Donnell MB, Cascio CN, Tinney F, Kang Y, Lieberman MD, Taylor SE, An L, Resnicow K, Strecher VJ. Self-affirmation alters the brain's response to health messages and subsequent behavior change. Proc Natl Acad Sci U S A. 2015 Feb 17;112(7):1977-82. doi: 10.1073/pnas.1500247112. Epub 2015 Feb 2. PMID 25646442
- [Background] Cascio CN, Carp J, O'Donnell MB, Tinney FJ Jr, Bingham CR, Shope JT, Ouimet MC, Pradhan AK, Simons-Morton BG, Falk EB. Buffering social influence: neural correlates of response inhibition predict driving safety in the presence of a peer. J Cogn Neurosci. 2015 Jan;27(1):83-95. doi: 10.1162/jocn_a_00693. PMID 25100217
- [Background] Kelly MP, Kriznik NM, Kinmonth AL, Fletcher PC. The brain, self and society: a social-neuroscience model of predictive processing. Soc Neurosci. 2019 Jun;14(3):266-276. doi: 10.1080/17470919.2018.1471003. Epub 2018 May 10. PMID 29718764
- [Background] Berkman ET, Falk EB. Beyond Brain Mapping: Using Neural Measures to Predict Real-World Outcomes. Curr Dir Psychol Sci. 2013 Feb;22(1):45-50. doi: 10.1177/0963721412469394. PMID 24478540
- [Background] Berkman ET, Falk EB, Lieberman MD. In the trenches of real-world self-control: neural correlates of breaking the link between craving and smoking. Psychol Sci. 2011 Apr;22(4):498-506. doi: 10.1177/0956797611400918. Epub 2011 Mar 4. PMID 21378368
- [Background] Kang Y, O'Donnell MB, Strecher VJ, Falk EB. Dispositional Mindfulness Predicts Adaptive Affective Responses to Health Messages and Increased Exercise Motivation. Mindfulness (N Y). 2017 Apr;8(2):387-397. doi: 10.1007/s12671-016-0608-7. Epub 2016 Sep 13. PMID 28344683
- [Background] Falk EB, Morelli SA, Welborn BL, Dambacher K, Lieberman MD. Creating buzz: the neural correlates of effective message propagation. Psychol Sci. 2013 Jul 1;24(7):1234-42. doi: 10.1177/0956797612474670. Epub 2013 May 30. PMID 23722983
- [Background] Lopez RB, Chen PA, Huckins JF, Hofmann W, Kelley WM, Heatherton TF. A balance of activity in brain control and reward systems predicts self-regulatory outcomes. Soc Cogn Affect Neurosci. 2017 May 1;12(5):832-838. doi: 10.1093/scan/nsx004. PMID 28158874
- [Background] Falk EB, Cascio CN, O'Donnell MB, Carp J, Tinney FJ Jr, Bingham CR, Shope JT, Ouimet MC, Pradhan AK, Simons-Morton BG. Neural responses to exclusion predict susceptibility to social influence. J Adolesc Health. 2014 May;54(5 Suppl):S22-31. doi: 10.1016/j.jadohealth.2013.12.035. PMID 24759437
- [Background] Brewer JA, Worhunsky PD, Carroll KM, Rounsaville BJ, Potenza MN. Pretreatment brain activation during stroop task is associated with outcomes in cocaine-dependent patients. Biol Psychiatry. 2008 Dec 1;64(11):998-1004. doi: 10.1016/j.biopsych.2008.05.024. Epub 2008 Jul 17. PMID 18635157
- [Background] Kosten TR, Scanley BE, Tucker KA, Oliveto A, Prince C, Sinha R, Potenza MN, Skudlarski P, Wexler BE. Cue-induced brain activity changes and relapse in cocaine-dependent patients. Neuropsychopharmacology. 2006 Mar;31(3):644-50. doi: 10.1038/sj.npp.1300851. PMID 16123763
- [Background] Paulus MP, Tapert SF, Schuckit MA. Neural activation patterns of methamphetamine-dependent subjects during decision making predict relapse. Arch Gen Psychiatry. 2005 Jul;62(7):761-8. doi: 10.1001/archpsyc.62.7.761. PMID 15997017
- [Background] Chua HF, Ho SS, Jasinska AJ, Polk TA, Welsh RC, Liberzon I, Strecher VJ. Self-related neural response to tailored smoking-cessation messages predicts quitting. Nat Neurosci. 2011 Apr;14(4):426-7. doi: 10.1038/nn.2761. Epub 2011 Feb 27. PMID 21358641
- [Background] Baek EC, Scholz C, O'Donnell MB, Falk EB. The Value of Sharing Information: A Neural Account of Information Transmission. Psychol Sci. 2017 Jul;28(7):851-861. doi: 10.1177/0956797617695073. Epub 2017 May 15. PMID 28504911
- [Background] Shadel WG, Martino SC, Setodji CM, Scharf DM, Kusuke D, Sicker A, Gong M. Hiding the tobacco power wall reduces cigarette smoking risk in adolescents: using an experimental convenience store to assess tobacco regulatory options at retail point-of-sale. Tob Control. 2015 Nov 23:tobaccocontrol-2015-052529 10.1136/tobaccocontrol-2015-052529. doi: 10.1136/tobaccocontrol-2015-052529. Online ahead of print. PMID 26598502
- [Background] Mendez D, Alshanqeety O, Warner KE. The potential impact of smoking control policies on future global smoking trends. Tob Control. 2013 Jan;22(1):46-51. doi: 10.1136/tobaccocontrol-2011-050147. Epub 2012 Apr 25. PMID 22535364
- [Background] Jamal A, King BA, Neff LJ, Whitmill J, Babb SD, Graffunder CM. Current Cigarette Smoking Among Adults - United States, 2005-2015. MMWR Morb Mortal Wkly Rep. 2016 Nov 11;65(44):1205-1211. doi: 10.15585/mmwr.mm6544a2. PMID 27832052
- [Background] Lee JG, Henriksen L, Rose SW, Moreland-Russell S, Ribisl KM. A Systematic Review of Neighborhood Disparities in Point-of-Sale Tobacco Marketing. Am J Public Health. 2015 Sep;105(9):e8-18. doi: 10.2105/AJPH.2015.302777. Epub 2015 Jul 16. PMID 26180986
- [Background] Klucharev V, Smidts A, Fernandez G. Brain mechanisms of persuasion: how 'expert power' modulates memory and attitudes. Soc Cogn Affect Neurosci. 2008 Dec;3(4):353-66. doi: 10.1093/scan/nsn022. Epub 2008 Aug 7. PMID 19015077
- [Background] Donny EC, Hatsukami DK. Randomized Trial of Reduced-Nicotine Standards for Cigarettes. N Engl J Med. 2016 Jan 28;374(4):396-7. doi: 10.1056/NEJMc1513886. No abstract available. PMID 26816022
- [Background] Mercincavage M, Souprountchouk V, Tang KZ, Dumont RL, Wileyto EP, Carmella SG, Hecht SS, Strasser AA. A Randomized Controlled Trial of Progressively Reduced Nicotine Content Cigarettes on Smoking Behaviors, Biomarkers of Exposure, and Subjective Ratings. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1125-33. doi: 10.1158/1055-9965.EPI-15-1088. Epub 2016 Apr 27. PMID 27197288
- [Background] Lochbuehler K, Mercincavage M, Tang KZ, Dana Tomlin C, Cappella JN, Strasser AA. Effect of message congruency on attention and recall in pictorial health warning labels. Tob Control. 2017 May 16:tobaccocontrol-2016-053615. doi: 10.1136/tobaccocontrol-2016-053615. Online ahead of print. PMID 28512171
- [Background] Strasser AA, Ashare RL, Kaufman M, Tang KZ, Mesaros AC, Blair IA. The effect of menthol on cigarette smoking behaviors, biomarkers and subjective responses. Cancer Epidemiol Biomarkers Prev. 2013 Mar;22(3):382-9. doi: 10.1158/1055-9965.EPI-12-1097. Epub 2013 Jan 18. PMID 23334588
- [Background] Barnett I, Onnela JP. Inferring mobility measures from GPS traces with missing data. Biostatistics. 2020 Apr 1;21(2):e98-e112. doi: 10.1093/biostatistics/kxy059. PMID 30371736
- [Background] Barnett I, Torous J, Staples P, Sandoval L, Keshavan M, Onnela JP. Relapse prediction in schizophrenia through digital phenotyping: a pilot study. Neuropsychopharmacology. 2018 Jul;43(8):1660-1666. doi: 10.1038/s41386-018-0030-z. Epub 2018 Feb 22. PMID 29511333
- [Background] Lee JG, Henriksen L, Myers AE, Dauphinee AL, Ribisl KM. A systematic review of store audit methods for assessing tobacco marketing and products at the point of sale. Tob Control. 2014 Mar;23(2):98-106. doi: 10.1136/tobaccocontrol-2012-050807. Epub 2013 Jan 15. PMID 23322313
- [Background] Whalen CK, Jamner LD, Henker B, Delfino RJ. Smoking and moods in adolescents with depressive and aggressive dispositions: evidence from surveys and electronic diaries. Health Psychol. 2001 Mar;20(2):99-111. PMID 11315734
- [Background] Pearson JL, Smiley SL, Rubin LF, Anesetti-Rothermel A, Elmasry H, Davis M, DeAtley T, Harvey E, Kirchner T, Abrams DB. The Moment Study: protocol for a mixed method observational cohort study of the Alternative Nicotine Delivery Systems (ANDS) initiation process among adult cigarette smokers. BMJ Open. 2016 Apr 22;6(4):e011717. doi: 10.1136/bmjopen-2016-011717. PMID 27105716
- [Background] Tseng TY, Ostroff JS, Campo A, Gerard M, Kirchner T, Rotrosen J, Shelley D. A Randomized Trial Comparing the Effect of Nicotine Versus Placebo Electronic Cigarettes on Smoking Reduction Among Young Adult Smokers. Nicotine Tob Res. 2016 Oct;18(10):1937-1943. doi: 10.1093/ntr/ntw017. Epub 2016 Jan 17. PMID 26783292
- [Background] Duncan DT, Kapadia F, Kirchner TR, Goedel WC, Brady WJ, Halkitis PN. Acceptability of Ecological Momentary Assessment Among Young Men Who Have Sex with Men. J LGBT Youth. 2017;14(4):436-444. doi: 10.1080/19361653.2017.1365038. Epub 2017 Sep 1. PMID 29988981
- [Background] Mead EL, Johnson SL, Siddiqui J, Butler J 3rd, Kirchner T, Feldman RH. Beyond blunts: Reasons for cigarette and cigar use among African American young adult dual users. Addict Res Theory. 2018;26(5):349-360. doi: 10.1080/16066359.2017.1366456. Epub 2017 Sep 1. PMID 30344466
- [Background] Chen-Sankey JC, Choi K, Kirchner TR, Feldman RH, Butler J 3rd, Mead EL. Flavored cigar smoking among African American young adult dual users: An ecological momentary assessment. Drug Alcohol Depend. 2019 Mar 1;196:79-85. doi: 10.1016/j.drugalcdep.2018.12.020. Epub 2019 Jan 31. PMID 30754022
- [Background] Vu M, Getachew B, Payne JB, Kirchner TR, Berg CJ. Initiation, continuation of use and cessation of alternative tobacco products among young adults: A qualitative study. Tob Prev Cessat. 2018 Feb;4:8. doi: 10.18332/tpc/84869. PMID 30272039
- [Background] Berg CJ, Haardorfer R, Payne JB, Getachew B, Vu M, Guttentag A, Kirchner TR. Ecological momentary assessment of various tobacco product use among young adults. Addict Behav. 2019 May;92:38-46. doi: 10.1016/j.addbeh.2018.12.014. Epub 2018 Dec 11. PMID 30579116
- [Background] Henriksen L, Feighery EC, Wang Y, Fortmann SP. Association of retail tobacco marketing with adolescent smoking. Am J Public Health. 2004 Dec;94(12):2081-3. doi: 10.2105/ajph.94.12.2081. PMID 15569957
- [Background] Roberts NJ, Kerr SM, Smith SM. Behavioral interventions associated with smoking cessation in the treatment of tobacco use. Health Serv Insights. 2013 Aug 11;6:79-85. doi: 10.4137/HSI.S11092. eCollection 2013. PMID 25114563
- [Background] Strasser AA, Tang KZ, Romer D, Jepson C, Cappella JN. Graphic warning labels in cigarette advertisements: recall and viewing patterns. Am J Prev Med. 2012 Jul;43(1):41-7. doi: 10.1016/j.amepre.2012.02.026. PMID 22704744
- [Background] Falk EB, Hyde LW, Mitchell C, Faul J, Gonzalez R, Heitzeg MM, Keating DP, Langa KM, Martz ME, Maslowsky J, Morrison FJ, Noll DC, Patrick ME, Pfeffer FT, Reuter-Lorenz PA, Thomason ME, Davis-Kean P, Monk CS, Schulenberg J. What is a representative brain? Neuroscience meets population science. Proc Natl Acad Sci U S A. 2013 Oct 29;110(44):17615-22. doi: 10.1073/pnas.1310134110. Epub 2013 Oct 22. PMID 24151336
- [Background] Cooper N, Tompson S, O'Donnell MB, Vettel JM, Bassett DS, Falk EB. Associations between coherent neural activity in the brain's value system during antismoking messages and reductions in smoking. Health Psychol. 2018 Apr;37(4):375-384. doi: 10.1037/hea0000574. Epub 2018 Feb 15. PMID 29446965
- [Background] Dore BP, Cooper N, Scholz C, O'Donnell MB, Falk EB. Cognitive regulation of ventromedial prefrontal activity evokes lasting change in the perceived self-relevance of persuasive messaging. Hum Brain Mapp. 2019 Jun 15;40(9):2571-2580. doi: 10.1002/hbm.24545. Epub 2019 Feb 17. PMID 30773729
- [Background] Kang Y, Cooper N, Pandey P, Scholz C, O'Donnell MB, Lieberman MD, Taylor SE, Strecher VJ, Dal Cin S, Konrath S, Polk TA, Resnicow K, An L, Falk EB. Effects of self-transcendence on neural responses to persuasive messages and health behavior change. Proc Natl Acad Sci U S A. 2018 Oct 2;115(40):9974-9979. doi: 10.1073/pnas.1805573115. Epub 2018 Sep 17. PMID 30224461
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Poldrack RA, Baker CI, Durnez J, Gorgolewski KJ, Matthews PM, Munafo MR, Nichols TE, Poline JB, Vul E, Yarkoni T. Scanning the horizon: towards transparent and reproducible neuroimaging research. Nat Rev Neurosci. 2017 Feb;18(2):115-126. doi: 10.1038/nrn.2016.167. Epub 2017 Jan 5. PMID 28053326
- [Background] Janes AC, Frederick Bd, Richardt S, Burbridge C, Merlo-Pich E, Renshaw PF, Evins AE, Fava M, Kaufman MJ. Brain fMRI reactivity to smoking-related images before and during extended smoking abstinence. Exp Clin Psychopharmacol. 2009 Dec;17(6):365-73. doi: 10.1037/a0017797. PMID 19968401
- [Background] Goudriaan AE, de Ruiter MB, van den Brink W, Oosterlaan J, Veltman DJ. Brain activation patterns associated with cue reactivity and craving in abstinent problem gamblers, heavy smokers and healthy controls: an fMRI study. Addict Biol. 2010 Oct;15(4):491-503. doi: 10.1111/j.1369-1600.2010.00242.x. Epub 2010 Sep 14. PMID 20840335
- [Background] Shiffman S, West R, Gilbert D; SRNT Work Group on the Assessment of Craving and Withdrawal in Clinical Trials. Recommendation for the assessment of tobacco craving and withdrawal in smoking cessation trials. Nicotine Tob Res. 2004 Aug;6(4):599-614. doi: 10.1080/14622200410001734067. PMID 15370156
- [Background] Sayette MA, Shiffman S, Tiffany ST, Niaura RS, Martin CS, Shadel WG. The measurement of drug craving. Addiction. 2000 Aug;95 Suppl 2(Suppl 2):S189-210. doi: 10.1080/09652140050111762. PMID 11002914
- [Background] Dunbar MS, Scharf D, Kirchner T, Shiffman S. Do smokers crave cigarettes in some smoking situations more than others? Situational correlates of craving when smoking. Nicotine Tob Res. 2010 Mar;12(3):226-34. doi: 10.1093/ntr/ntp198. Epub 2010 Feb 4. PMID 20133379
- [Background] Mooney M, Green C, Hatsukami D. Nicotine self-administration: cigarette versus nicotine gum diurnal topography. Hum Psychopharmacol. 2006 Dec;21(8):539-48. doi: 10.1002/hup.808. PMID 17066490
- [Background] Benowitz NL, Kuyt F, Jacob P 3rd. Circadian blood nicotine concentrations during cigarette smoking. Clin Pharmacol Ther. 1982 Dec;32(6):758-64. doi: 10.1038/clpt.1982.233. PMID 7140139
- [Background] Groefsema M, Engels R, Luijten M. The role of social stimuli content in neuroimaging studies investigating alcohol cue-reactivity. Addict Behav. 2016 Jul;58:123-8. doi: 10.1016/j.addbeh.2016.02.033. Epub 2016 Feb 17. PMID 26922160
- [Background] Drummond DC. What does cue-reactivity have to offer clinical research? Addiction. 2000 Aug;95 Suppl 2:S129-44. doi: 10.1080/09652140050111708. PMID 11002908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults who smoked cigarettes daily were recruited across PA, DE, and NJ to complete a multi-part, remote study. Recruitment materials for this study were primarily distributed by a clinical trials recruitment company, which utilized study advertisements to engage participants on digital platforms such as Facebook, Google, and WebMD. All recruitment materials included links directing potential participants to the initial screening survey.
Pre-assignment Details: Participants completed several screening steps to confirm eligibility and interest in the study. If eligible, they completed the first online survey session, and then began the baseline period, during which they answered questions about their cigarette craving and smoking multiple times daily and recorded their geolocation through the Google Maps smartphone application. Participants who completed the baseline period and began the intervention period were assigned to an experimental condition.
Groups:
- Unassigned: Participants who enrolled in the study but did not complete the baseline period and therefore were not assigned an experimental condition
Period: Baseline Period
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control | Unassigned
Started (Consented to participate) | 109 | 109 | 76 | 49
Began Baseline Period | 109 | 109 | 76 | 36
Completed | 109 | 109 | 76 | 10
Not Completed | 0 | 0 | 0 | 39
Period: Intervention Period
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control | Unassigned
Started | 109 | 109 | 76 | 0 (Not all participants who completed the baseline period began the intervention period (more specifically, the 10 participants who completed baseline but did not begin the intervention are classed as "unassigned").)
Completed All Store Visits (Participants could complete the final study session without having completed the full intervention of making 20 visits to their assigned store.) | 55 | 46 | 0 (Participants in the control condition did not make store visits as part of the protocol) | 0
Completed | 88 | 92 | 74 | 0
Not Completed | 21 | 17 | 2 | 0
Period: fMRI Scans
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control | Unassigned
Started | 10 | 13 | 13 | 1
Completed Second Scan (The original version of the study protocol required 2 fMRI scan sessions, one prior to the intervention period and one after the intervention period. We changed the study protocol during the COVID-19 pandemic to make fMRI scans optional, and to only offer a single scan session after the intervention period.) | 1 | 3 | 5 | 0
Completed | 10 | 12 | 13 | 0
Not Completed | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population includes each individual who signed the informed consent form.
Groups:
- Unassigned: Participants who enrolled in the study, but did not complete the baseline period and were therefore not assigned to an experimental condition
- Total: Total of all reporting groups
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control | Unassigned | Total
Number analyzed (Participants) | 109 | 109 | 76 | 49 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 42 (11) | 42 (10) | 43 (11) | 43 (11)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/gender: Female | 59 | 60 | 42 | 20 | 181
  Sex/gender: Male | 46 | 44 | 32 | 25 | 147
  Sex/gender: Other | 3 | 5 | 1 | 0 | 9
  Sex/gender: Unknown | 1 | 0 | 1 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 3 | 3 | 22
  Not Hispanic or Latino | 99 | 102 | 71 | 42 | 314
  Unknown or Not Reported | 1 | 0 | 2 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 3 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 27 | 24 | 17 | 25 | 93
  White | 75 | 69 | 47 | 17 | 208
  More than one race | 2 | 9 | 4 | 0 | 15
  Unknown or Not Reported | 4 | 4 | 4 | 5 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 109 | 109 | 76 | 49 | 343
Daily cigarette craving [Mean (Standard Deviation); unit: units on a scale] — Participants were asked 4 times per day, for the 14 days of the baseline period, to rate their level of craving for a cigarette. They responded to the question "Right now, how much do you want to smoke a cigarette?" using a 100-point scale from 0 (not at all) to 100 (extremely). Craving ratings were first averaged within each day, for each participant; then were averaged across the baseline period days for each participant; and finally averaged across participants in each group. Population: Some participants in the Unassigned group did not respond to any daily messages and are not represented in the average.
  units on a scale
    number analyzed (Participants) | 109 | 109 | 76 | 28 | 322
    (all) | 47.89 (20.70) | 49.17 (19.61) | 48.03 (20.81) | 59.86 (19.42) | 49.40 (20.43)
Daily cigarette count [Mean (Standard Deviation); unit: cigarettes] — Participants were asked 2 times per day, for each day of the 14 day baseline period, to respond to the question, "Within [timeframe], how many cigarettes did you smoke?". We calculated a daily sum for each individual, imputing missing counts from the average of that individual's prior reports (missing values for the first daily survey were imputed from the average of that participant's first daily survey answers; and vice versa for the second survey). We averaged the daily counts for each participant, and then averaged across participants. Population: Some participants in the Unassigned group did not respond to any daily messages and are not represented in the average.
  cigarettes
    number analyzed (Participants) | 109 | 109 | 76 | 28 | 322
    (all) | 13.29 (6.35) | 14.17 (19.18) | 14.05 (9.84) | 14.17 (9.18) | 13.71 (8.71)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Cigarette Craving During the Experimental Manipulation Period
Description: Participants were asked 4 times per day, for the 28 days of the intervention period, to rate their level of craving for a cigarette. They responded to the question "Right now, how much do you want to smoke a cigarette?" using a 100-point scale from 0 (not at all) to 100 (extremely). Craving ratings were first averaged within each day, for each participant; then were averaged across the intervention period days for each participant; and finally averaged across participants in each group.
Time Frame: 4-week experimental manipulation period
Population: All participants who responded to any craving rating questions during the intervention period are included in this average. Participants in the "unassigned" group did not begin the intervention period and therefore are have no outcome data to report.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control
Number analyzed (Participants) | 101 | 104 | 75
units on a scale | 48.33 (25.30) | 49.14 (22.96) | 47.17 (24.24)
Statistical Analysis 1: Comparison: Tobacco Retailer Group vs Non-tobacco Retailer Group; Our hypothesis was that craving would be higher for those in the Tobacco retailer group, relative to the Nontobacco retailer group, during the intervention phase but not the baseline phase. We tested the interaction between study phase and experimental condition, in a model where the baseline was the reference study phase and Tobacco group was the reference experimental condition; Test type: Superiority — Linear mixed effects; p = 0.74, Mixed Models Analysis — Statistical significance was evaluated at α = 0.05; Slope = -0.64, Standard Error of Mean 1.95
Statistical Analysis 2: Comparison: Tobacco Retailer Group vs Control; Our hypothesis was that craving would be higher for those in the Tobacco retailer group, relative to the control group, during the intervention phase but not the baseline phase. We tested the interaction between study phase and experimental condition, in a model where the baseline was the reference study phase and Tobacco group was the reference experimental condition; Test type: Superiority — Linear mixed effects; p = 0.69, Mixed Models Analysis — Statistical significance was evaluated at α = 0.05; Slope = -0.84, Standard Error of Mean 2.12

2. Primary Outcome: Self-reported Number of Cigarettes Smoked Per Day During the Experimental Manipulation Period
Description: Participants were asked 2 times per day, for the 28 days of the intervention period, to respond to the question, "Within [timeframe], how many cigarettes did you smoke?". We calculated a daily sum for each individual, imputing missing counts from the average of that individual's prior reports (missing values for the first daily survey were imputed from the average of that participant's first daily survey answers; and vice versa for the second survey). We averaged the daily counts for each participant, and then averaged across participants.
Time Frame: 4-week experimental manipulation period
Population: All participants who responded to any cigarette consumption questions during the intervention period are included in this average. Participants in the "unassigned" group did not begin the intervention period and therefore are have no outcome data to report.
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control
Number analyzed (Participants) | 101 | 104 | 75
cigarettes | 12.72 (6.26) | 12.88 (8.27) | 13.64 (7.55)
Statistical Analysis 1: Comparison: Tobacco Retailer Group vs Non-tobacco Retailer Group; Our hypothesis was that cigarettes smoked would be higher for those in the Tobacco retailer group, relative to the Nontobacco retailer group, during the intervention phase but not the baseline phase. We tested the interaction between study phase and experimental condition, in a model where the baseline was the reference study phase and Tobacco group was the reference experimental condition; Test type: Superiority — Linear mixed effects; p = 0.49, Mixed Models Analysis — Statistical significance was evaluated at α = 0.05; Slope = -0.37, Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Tobacco Retailer Group vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — Linear mixed effects; p = 0.72, Mixed Models Analysis — Statistical significance was evaluated at α = 0.05; Slope = 0.21, Standard Error of Mean 0.59

3. Primary Outcome: Brain Activity (Measured by Functional Magnetic Resonance Imaging) in a Priori Regions of Interest, in Response to Standardized Smoking vs Nonsmoking Cues.
Description: In key neural cue reactivity regions (based on prior work), we extracted estimates of neural activity during exposure to standardized smoking cues (e.g., photographs of a cigarette pack) and during exposure to standardized nonsmoking cues (approximately compositionally matched, e.g., a pack of pencils). We used SPM12 to create first-level (within-subject) linear regression models to estimate BOLD (blood oxygenation level dependent) activity at each voxel across all repetitions of each task condition, within each subject; and to create contrast estimates comparing task conditions. We used nilearn tools to average task condition contrast estimates across voxels within the regions of interest for each participant. The data values below reflect this contrast estimate - the difference in neural activity as percent change in BOLD signal between the standardized smoking cues condition and the standardized nonsmoking cues condition.
Time Frame: [Time Frame: For 822815, fMRI scan 1 (at least 2 weeks after initial enrollment); for 850796, fMRI scan 1 (at least 6 weeks after initial enrollment)]]
Population: Participants who completed at least one scan and whose data passed quality thresholds for in-scanner movement and response rate. Due to COVID-19 pandemic restrictions during data collection, we changed the protocol to make the fMRI scan optional, which means that we do not have adequate statistical power to test experimental group differences. No participants in the "unassigned" group were scanned, since they did not begin the intervention period.
Measure: Mean (Standard Deviation); unit: percent change in BOLD signal
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control
Number analyzed (Participants) | 7 | 10 | 11
percent change in BOLD signal | 0.021 (0.089) | -0.025 (0.080) | 0.035 (0.120)

4. Primary Outcome: Brain Activity (Measured by fMRI), in a Priori Regions of Interest, in Response to Retail Smoking vs Nonsmoking Cues
Description: In key neural cue reactivity regions (based on prior work), we will extract estimates of neural activity during exposure to images showing the cash register area at a convenience store which sells tobacco products, and has tobacco products and tobacco marketing on display behind the register (the "power wall"; tobacco retail images), and during exposure to nonsmoking cues. We used SPM12 to create first-level (within-subject) linear regression models to estimate BOLD (blood oxygenation level dependent) activity at each voxel across all repetitions of each task condition, within each subject; and to create contrast estimates comparing task conditions. We used nilearn tools to average task condition contrast estimates across voxels within the regions of interest for each participant. The data values below reflect this contrast estimate - the difference in neural activity as percent change in BOLD signal between the retail smoking cues condition and the nonsmoking cues condition.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change in BOLD signal
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control
Number analyzed (Participants) | 7 | 10 | 11
percent change in BOLD signal | 0.062 (0.118) | 0.012 (0.092) | 0.018 (0.108)

ADVERSE EVENTS:
Time Frame: Period of enrollment for each participant (approximately 6 weeks)
Groups:
- Unassigned: Participants who began the baseline period, but did not begin the intervention period and therefore were not assigned to an experimental group.
Arm/Group | Tobacco Retailer Group | Non-tobacco Retailer Group | Control | Unassigned
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/109 | 0/76 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/109 | 5/109 | 0/76 | 0/49
Other Adverse Events (participants affected / at risk) | 0/109 | 0/109 | 0/76 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tobacco Retailer Group (N=109) | Non-tobacco Retailer Group (N=109) | Control (N=76) | Unassigned (N=49)
Hospitalization (General disorders) | 2 | 5 | 0 | NA — All hospitalizations were unrelated to participation in the study

LIMITATIONS AND CAVEATS:
Due to COVID-19 pandemic-related constraints and delays, we were unable to reach our goal of 60 complete datasets per condition. We prioritized remote participation and made fMRI scans optional. This resulted in few participants completing fMRI scans. Our planned analyses investigating the effects of intervention group assignment on smoking and craving are well-powered with this sample size, but examination of intervention effects on neural responses to tobacco marketing is not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT04279483/Prot_SAP_000.pdf
  • Informed Consent Form: fMRIconsent (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04279483/ICF_001.pdf
  • Informed Consent Form: ScreeningConsent (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT04279483/ICF_002.pdf
  • Informed Consent Form: MainConsent (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT04279483/ICF_003.pdf
  • Informed Consent Form: fMRIScreenConsent (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT04279483/ICF_004.pdf